CLINICAL TRIAL: NCT06996925
Title: Erectile Dysfunction and the Mind: Evaluating the Influence of Depression and Illness Beliefs on Treatment Progression
Brief Title: Depression, Illness Perception, and Erectile Dysfunction Outcomes
Status: Enrolling by invitation | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nazım Furkan Günay, Urology specialist, Haseki Training and Research Hospital
Other Study IDs: 19.03.2025/23-2025
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Erectile Dysfunction; Depression; Perception and Beliefs
Keywords: erectile dysfunction; Depression; self perception
MeSH Terms: conditions — Erectile Dysfunction; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Erectile Dysfunction: This study includes adult male participants aged 18 and older who have been clinically diagnosed with erectile dysfunction (ED). All participants will have the condition of interest (ED), and there is no control group without the condition. The study group is homogeneous in that it consists solely of patients with ED, allowing for the evaluation of intra-individual changes over time in illness perception, depressive symptoms, and erectile functio

SUMMARY:
The goal of this observational study is to evaluate the impact of illness perception and depressive symptoms on treatment outcomes in adult male patients diagnosed with erectile dysfunction (ED).

The main questions it aims to answer are:

Is there a relationship between negative illness perception and increased severity of depressive symptoms in ED patients? Does the change in illness perception over time correlate with changes in erectile function and depression levels?

Participants will:

Complete the IIEF-5 (International Index of Erectile Function - 5) to assess erectile dysfunction severity, Complete the B-IPQ (Brief Illness Perception Questionnaire) to evaluate their cognitive and emotional representations of ED, Complete the PHQ-9 (Patient Health Questionnaire - 9) to measure depressive symptoms, Repeat these assessments at baseline and at a 1-month follow-up. This study does not involve any intervention or comparison group. It is designed to track psychological and clinical changes over time and explore modifiable psychological predictors in the management of ED.

DETAILED DESCRIPTION:
This prospective, observational study aims to investigate the relationship between illness perception and depressive symptoms in patients diagnosed with erectile dysfunction (ED), and how these factors influence treatment response over time. Erectile dysfunction is a multifactorial condition that significantly affects quality of life and can be shaped by psychological and cognitive factors, including patients' perceptions of their disease.

A total of 120 adult male participants (aged >18 years) diagnosed with ED will be enrolled from multiple urology centers. Patients will complete three validated instruments at baseline and again at a 1-month follow-up:

IIEF-5 (International Index of Erectile Function - 5): to assess severity of erectile dysfunction.

B-IPQ (Brief Illness Perception Questionnaire): to evaluate cognitive and emotional representations of their condition.

PHQ-9 (Patient Health Questionnaire - 9): to screen for and quantify depressive symptoms.

The primary outcome of the study is to determine the association between baseline illness perception (as measured by B-IPQ) and the severity of depressive symptoms (PHQ-9 scores). Secondary outcomes include changes in erectile function (IIEF-5) and depressive symptoms at 1 month, and whether these changes correlate with changes in illness perception. Additionally, specific components of illness perception such as personal control, treatment control, concern, and emotional response will be analyzed in relation to treatment adherence and psychological well-being.

Data Quality and Management Procedures:

A structured case report form (CRF) will be used for consistent data entry. A data dictionary will define each variable and ensure uniform interpretation of collected data.

Data checks will be performed to validate internal consistency (e.g., checking for missing or out-of-range values).

Source data verification will involve comparison of collected responses with patients' medical records when applicable.

Standard Operating Procedures (SOPs) will be followed for data collection, participant follow-up, and data management.

Sample Size and Statistical Plan:

A power analysis indicated a required sample size of 120 participants to detect a moderate correlation (r = 0.3) between illness perception and depressive symptoms with 80% power and a 5% significance level.

Statistical analysis will include:

Descriptive statistics for demographic and clinical variables. Pearson or Spearman correlation analysis between B-IPQ, PHQ-9, and IIEF-5 scores.

Paired t-tests or Wilcoxon signed-rank tests to assess within-group changes over time.

Multivariate regression analysis to control for potential confounders such as age, comorbidities, and duration of ED.

Missing Data Plan:

Cases with missing responses will be addressed using multiple imputation methods where appropriate. Sensitivity analyses will be conducted to assess the impact of missing data on study outcomes.

This study will provide insight into how modifiable psychological factors such as illness beliefs influence both psychological distress and sexual health, potentially informing future patient education and intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years or older
* Diagnosed with erectile dysfunction by a physician
* Able and willing to provide written informed consent

Exclusion Criteria:

* History of severe psychiatric disorders (e.g., schizophrenia, bipolar disorder)
* Ongoing or prior hormonal therapy or active cancer treatment
* Neurological conditions that could impact erectile function

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the outpatient urology clinics of Haseki Training and Research Hospital and collaborating centers. All participants will be adult male patients who present with complaints consistent with erectile dysfunction and meet the diagnostic criteria during clinical evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Association between illness perception and depressive symptoms | Baseline and 1-month follow-up
  Change in depressive symptom scores (Patient Health Questionnaire-9, PHQ-9; range 0-27; higher scores indicate worse depressive symptoms) in relation to illness perception scores (Brief Illness Perception Questionnaire, B-IPQ; range 0-80; higher scores indicate more negative illness perceptions) at baseline and 1-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Furkan Gunay, Medical doctor, Principal Investigator — Haseki Education and Research Hospital
Locations (1):
- Haseki Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available to qualified researchers upon reasonable request. Requests will be evaluated by the principal investigator to ensure that the proposed use is scientifically and ethically appropriate. Data will be shared under a formal data use agreement that protects participant confidentiality and complies with ethical standards.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available starting 6 months after publication of the study results and will remain available for up to 2 years.
Access Criteria: Qualified researchers affiliated with academic institutions, research organizations, or healthcare institutions may request access to the data.
  What information they can access:
  * Individual participant data (IPD)
  * Study protocol
  * Statistical analysis plan
  * Informed consent form (upon request)
  How they can access it:
  Researchers must submit a formal request to the principal investigator including a brief research proposal and institutional ethical approval. If the request is approved, a data use agreement (DUA) must be signed to ensure appropriate data handling and confidentiality. Access will then be granted through a secure, password-protected electronic transfer system managed by the study team.
URL: https://vivli.org

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT06996925/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT06996925/ICF_001.pdf